CLINICAL TRIAL: NCT00630409
Title: Phase II Clinical Trial of Gemcitabine and Doxil® for Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Leonard Appleman, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-033
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Kidney Cancer; Gemcitabine; Doxil; Chemotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Gemcitabine; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients will receive 3 cycles of therapy as an outpatient. Each 21-day cycle of therapy will comprise: Gemcitabine: IV on days 1 and 8. Doxil: on day 1. Patients with either responding or stable disease will continue to receive additional 3 cycles of therapy with gemcitabine and Doxil until there is radiological evidence of disease progression or they are unable or unwilling to continue treatment.
  Interventions: Drug: Gemcitabine; Drug: Doxil

INTERVENTIONS:
Drug: Gemcitabine — 800 mg IV day 1 and 8
  Other Names: Gemzar
Drug: Doxil — 24 mg/m2 every 21 days IV
  Other Names: doxorubicin; adriamycin

SUMMARY:
The purpose of this study is to test the hypothesis that the combination of gemcitabine and doxil will have clinical activity in patients with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Patients with metastatic renal cell carcinoma who have received prior therapy with sorafenib, sunitinib or temsirolimus and have progressive disease may participate in this study if all eligibility criteria are met. Doxil will be administered on day 1 and gemcitabine on day 1 and 8 of a 21 day cycle. Tumor responses will be evaluated by RECIST. Up to six cycles of study treatment may be administered. Cardiac ejection fraction will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal cell carcinoma who have had disease progression through sorafenib, sunitinib, or temsirolimus (within 6 months of treatment).
* Diagnosis of RCC has been confirmed by pathological or cytological examination of tissue obtained from the primary tumor or a metastatic site.
* Clear cell and non-clear cell histological variants are permitted.
* With the exception of prior gemcitabine or any anthracycline (e.g., doxorubicin, epirubicin, DOXIL), any number of prior therapies with are permitted.
* Prior nephrectomy is permitted but not required for eligibility.
* Patients who have received palliative radiation therapy (XRT) to any area other than the brain (see below) may begin therapy immediately after completion of XRT as long as the irradiated lesion(s) is/are not used for clinical response assessment.

Brain metastases:

* Patients requiring XRT or gamma-knife (or similar) therapy to the brain must wait at least 4 weeks after the completion of irradiation before starting therapy.
* Only patients with either stable or regressing brain metastases after irradiation, as determined by CT or MRI, are eligible for therapy.

  * No systemic therapy within 28 days prior to enrollment except as below:
  * No sorafenib, sunitinib, temsirolimus therapy within 14 days prior to enrollment.
  * Toxicities from prior therapy must have resolved to ≤Grade I.
  * Survival: anticipated survival of at least three months.
  * Renal function: creatinine ≥ 2.0 mg/dL.
* Patients must have a MUGA scan or 2-D echocardiogram indicating an ejection fraction of ≥50% within 42 days prior to the first dose of study drug. The method used at baseline must be used for later monitoring.
* Prior to each new cycle of therapy: hepatic function: AST, ALT ≥ 3X the upper limit of normal, unless the liver is involved by tumor, in which case the transaminases must be ≥ 5X the upper limit of normal. Total bilirubin must be ≥ 1.5 mg/dL.
* Prior to each new cycle of therapy: bone marrow function: absolute neutrophil count (ANC) ≥ 1,500; platelet count ≥ 100,000; hemoglobin ≥ 10 g/dL.
* Performance status: ECOG 0 or 1.
* Age: ≥ 18 years.
* Signed informed consent must be obtained from participating individuals.
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide, or surgical sterilization) during treatment and for three months after completing treatment. If a patient becomes pregnant while on study, the patient will be removed from the study and all drug treatment discontinued.

Exclusion Criteria:

* Patients who have received prior therapy with gemcitabine or an anthracycline drug (e.g., doxorubicin, epirubicin, DOXIL).
* Patients with untreated central nervous system metastases.
* Patients with active bacterial or fungal infections.
* Patients with psychiatric disorders that would interfere with consent, compliance with protocol requirements, or follow-up.
* Patients with a history of prior malignancy other than RCC, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
* Patients with any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for the entry into the study.
* Pregnant or lactating women.
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the component of DOXIL,
* History of cardiac disease with New York Heart Association Class II or greater cardiac function or clinical evidence of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV): Patients will receive 3 cycles of therapy as an outpatient. Each 21-day cycle of therapy will comprise: Gemcitabine: IV on days 1 and 8. Doxil: on day 1. Patients with either responding or stable disease will continue to receive additional 3 cycles of therapy with gemcitabine and Doxil until there is radiological evidence of disease progression or they are unable or unwilling to continue treatment.
  Gemcitabine: 800 mg IV day 1 and 8
  Doxil: 24 mg/m2 every 21 days IV
Period: Overall Study
Arm/Group | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV)
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV)
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 59 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Number of participants that experienced response/total number of participants per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan. Response was defined as Complete Response (CR), the disappearance of all target lesions; Partial Response (PR), a 30% or greater decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 18 weeks for individual; Up to 40 months for cohort
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV)
Number analyzed (Participants) | 5
percentage of participants | 0

2. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 40 months
Population: Due to lack of follow-up, objective could not be determined.
Measure: Median (95% Confidence Interval); unit: participants
Groups:
- Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV): Patients will receive 3 cycles of therapy as an outpatient. Each 21-day cycle of therapy will comprise: Gemcitabine: IV on days 1 and 8. Doxil: on day 1. Patients with either responding or stable disease will continue to receive additional 3 cycles of therapy with gemcitabine and Doxil until there is radiological evidence of disease progression or they are unable or unwilling to continue treatment.
  Gemcitabine: 800 mg IV day 1 and 8 + Doxil: 24 mg/m2 every 21 days IV
Arm/Group | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV)
Number analyzed (Participants) | 5
participants | NA [NA to NA] — Median time to progression was not reached due to lack of events; insufficient number of participants with events.

ADVERSE EVENTS:
Arm/Group | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV)
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine 800 mg/m^2 + Doxil 24 mg/m^2 (IV) (N=5)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (total WBC) (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Platelets (Investigations) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Rigors/chills (General disorders) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Injection site reaction/extravasation changes (General disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Creatinine (Investigations) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Neurology - Other (Nervous system disorders) | 2
Pain, Back (Musculoskeletal and connective tissue disorders) | 3
Pain, Joint (Musculoskeletal and connective tissue disorders) | 1
Pain, Liver (Hepatobiliary disorders) | 1
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes